CLINICAL TRIAL: NCT06737497
Title: Analysis of the Effectiveness and Safety of Retrograde Intrarenal Surgery (RIRS) Under Local Anesthesia and Its Influencing Factors
Brief Title: Analysis of the Effectiveness and Safety of RIRS Under Local Anesthesia and Its Influencing Factors
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Ph.D and M.D, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: Guohua Zeng
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-12

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: retrograde Intrarenal Surgery ( RIRS ) under local anesthesia — retrograde Intrarenal Surgery ( RIRS ) under local anesthesia

SUMMARY:
Retrograde intrarenal surgery (RIRS) is a well-established technique and is the first-line treatment option for upper urinary tract stones <2cm. Currently, most ureteroscopic procedures are performed under general or epidural anesthesia, both of which are safe and feasible. In recent years, more and more studies have shown that retrograde intrarenal surgery (RIRS) under local anesthesia is safe and feasible. However, we can see that the current studies on RIRS under local anesthesia are mostly case reports, and there is a lack of systematic studies on the safety and effectiveness of RIRS under local anesthesia and its influencing factors. Therefore, the researchers hope to conduct a single-center prospective observational study to explore the safety, effectiveness and influencing factors of RIRS under local anesthesia, so as to optimize the surgical process of RIRS under local anesthesia, improve the surgical success rate and ensure surgical safety。

ELIGIBILITY:
Inclusion Criteria:

1. Kidney stones or upper ureteral stones 1-4cm;
2. Age 18-70 years old;
3. American Society of Anesthesiologists(ASA) score Ⅰ, Ⅱ and Ⅲ;

Exclusion Criteria:

1. Surgical operations other than RIRS are required for patients with middle and lower ureteral calculi;
2. There are anatomical abnormalities, such as ureteral stenosis, urine flow diversion, ectopic kidney, horseshoe kidney, duplicate kidney, etc.
3. Severe heart, brain and lung diseases;
4. Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper urinary tract stones who are willing to undergo RIRS under local anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
pain score | 1 day after sugery
  Visual Analogue Scale(VAS)，The basic method is to use a moving ruler about 10cm long, with 10 scales on one side and "0" and "10" points on both ends, where 0 represents no pain and 10 represents the most unbearable pain.
Operative time | During surgery
  Surgery duration, minutes. From the insertion of the guide wire to the end of the indwelling ureteral stent.

SECONDARY OUTCOMES:
stone-free rate | From enrollment to the end of treatment at 1 month
  A low-dose and ultrathin 2-mm spiral CT was performed at 1 day postoperatively for evaluation of fnal SFR. Stone-free status was defined as no fragments observed or clinically insignifcant residual fragments (CIRF)<2 mm.
stone-free rate | From enrollment to the end of treatment at 24 hours
  A low-dose and ultrathin 2-mm spiral CT was performed at 1 day postoperatively for evaluation of fnal SFR. Stone-free status was defined as no fragments observed or clinically insignifcant residual fragments (CIRF)<2 mm.
Complication rate | 1 month after sugery
  Complication is defined as any adverse event occurred intraoperatively or ≤1 month postoperatively, including intraoperative bleeding, postoperative pain and so on.The investigator will invaluate perioperative complications by modified Clavien system

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China